CLINICAL TRIAL: NCT03814434
Title: Surgical Treatment of Periimplantitis in Patients With Risk Factors: Heavy Smokers, Type 2 Diabetic and Chronic Periodontitis Patients
Brief Title: Surgical Treatment of Periimplantitis in Patients With Risk Factors
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Luiz Antonio Pugliesi Alves de Lima (Other)
Responsible Party: Sponsor-Investigator, Luiz Antonio Pugliesi Alves de Lima, Associate Professor, University of Sao Paulo
Organization: University of Sao Paulo (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RiskFactorsSurgPeriimplantitis
Record Dates: First submitted 2019-01-21; First posted 2019-01-24 (Actual); Last update posted 2019-03-11 (Actual); Status verified 2019-03

CONDITIONS: Peri-Implantitis; Type 2 Diabetes Mellitus; Smoking, Cigarette; Periodontal Diseases
Keywords: peri-implantitis; inflammation; Therapy
MeSH Terms: conditions — Peri-Implantitis; Diabetes Mellitus, Type 2; Cigarette Smoking; Periodontal Diseases; Inflammation | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Intervention Model Description: This is not a randomized study. All patients will entered the study after being diagnosed with periimplantitis. Patients will be allocated to different groups according to their condition: Heavy Smokers, Type 2 Diabetes Mellitus, Chronic periodontitis and systemically healthy patients (control group).
Who Masked: Investigator, Outcomes Assessor
Masking Description: Surgeon will not be aware of group being treated. Analyses of the data and statistics will not show explain what group has originated the data. Groups will be identified as A, B, C or D.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Smokers with Periimplantitis group (Experimental): Heavy smokers patients with periimplantitis will be evaluated and will have their clinical, biological and radiographic data collected at baseline, after non-surgical and surgical treatment and after 3, 6 and 12 months.
  Interventions: Procedure: Non-Surgical treatment; Procedure: Surgical Treatment
- Type 2 Diabetes with Periimplantitis group (Experimental): Patients diagnosed with Type 2 Diabetes with periimplantitis will be evaluated and will have their clinical, biological and radiographic data collected at baseline, after non-surgical and surgical treatment and after 3, 6 and 12 months.
  Interventions: Procedure: Non-Surgical treatment; Procedure: Surgical Treatment
- Chronic Periodontitis with Periimplantitis group (Experimental): Patients diagnosed with Chronic Periodontitis and periimplantitis will be evaluated and will have their clinical, biological and radiographic data collected at baseline, after non-surgical and surgical treatment and after 3, 6 and 12 months.
  Interventions: Procedure: Non-Surgical treatment; Procedure: Surgical Treatment
- Control with Periimplantitis group (Experimental): Systemically healthy patients with periimplantitis will be included in this group. Patients will be evaluated and will have their clinical, biological and radiographic data collected at baseline, after non-surgical and surgical treatment and after 3, 6 and 12 months.
  Interventions: Procedure: Non-Surgical treatment; Procedure: Surgical Treatment

INTERVENTIONS:
Procedure: Non-Surgical treatment — Implant and teeth surfaces decontamination through scaling and planning, Curettage, profilaxys and Oral Hygiene orientation
Procedure: Surgical Treatment — Anaesthesia, Incision, curettage, Treatment of the contaminated implant surface, Irrigation with saline, Guided Bone Regeneration and suture

SUMMARY:
This study evaluates clinical and radiographic parameters among riks factor groups in patients with periimplantitis. This study will also treat and evaluate the patients response before and after surgical treatment.

DETAILED DESCRIPTION:
Periimplantitis (PI) is an inflammatory process that results in tissue attachment bone loss around the implant. Periodontal disease, smoke habit and type 2diabetes mellitus have been recognized as potential risk factor indicators that might lead to complications establishment and progression around dental implants. PI treatment predictability has been shown limited and influenced by factors not totally clarified. The aim of this study is to evaluate the reparative response after PI surgical treatment at clinical and radiographic levelsin risk factors patients: type 2 diabetes mellitus, smokers and chronic periodontal disease.

ELIGIBILITY:
Inclusion Criteria:

Implants diagnosed with peri-implantitis with boné defects; Probing depth ≥ 4mm; Positive Bleeding on Probing and Suppuration score; Radiographic Bone Loss ≥ 3mm; Generalized Chronic Periodontitis (Armitage, 1999); Heavy Smokers (> 10 cigarets per day); Type 2 Diabetes Mellitus tipo 2 (ADA, 2005) with HbA1c between 6.5% and 7.5%

Exclusion Criteria:

Complete Edentulism; Mucosal disease; Alcohol abuse; Systemic disease except type 2 Diabetes Mellitus, that might interfere in periimplantitis progression; Medication intake: anticoagulants, antineoplasics, contraceptives, bisphosphonates and antidepressives; Medication intake in the last 6 months: antibiotics; Medication intake in the last 3 months: antiinflammatories; Aggressive Periodontitis and Anaphylactic shock history; Periodontal treatment in the last 6 months before the baseline; Periodontal Pockets > 7mm; Light Smokers (< 10 cigarets/day); Implant Mobility.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-05-28 (Actual); Primary Completion 2020-01-28 (Estimated); Study Completion 2020-01-28 (Estimated)

PRIMARY OUTCOMES:
Radiographic Bone height Gain | 3 months
  Radiographic Bone Height Gain Comparison to baseline 3 months after surgical treatment

SECONDARY OUTCOMES:
Periimplant Pocket probing depth | 3 months
  Periimplant probing depth comparison to baseline 3 months after surgical treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Faculdade de Odontologia Universidade de Sao Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No